CLINICAL TRIAL: NCT02307825
Title: Azithromycin as add-on Therapy in Patients Failing Medical and Surgical Treatment for Chronic Rhinosinusitis: a Double-blind, Randomized, Placebo-controlled Trial
Brief Title: Azithromycin for Patients With Chronic Rhinosinusitis Failing Medical and Surgical Therapy
Acronym: AZI-CRS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14.140
Record Dates: First submitted 2014-11-11; First posted 2014-12-04 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2016-09

CONDITIONS: Chronic Rhinosinusitis; High-risk Patient
Keywords: Azithromycin; Endoscopic sinus surgery
MeSH Terms: interventions — Azithromycin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Azithromycin (Active Comparator): Patients will receive the active study drug, azithromycin, as well as sinus irrigations with budesonide.
  Interventions: Drug: Azithromycin
- Placebo (Placebo Comparator): Patients will receive a placebo as well as sinus irrigations with budesonide.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — The drug will be taken three times a week for four months.
  Other Names: Zithromax
  Arms: Azithromycin
Drug: Placebo — The placebo will be taken three times a week for four months.
  Other Names: No other name
  Arms: Placebo

SUMMARY:
Justification: Chronic rhinosinusitis (CRS) is one of the most common inflammatory diseases with an incidence and prevalence superior to 10%. Unfortunately, more than 30% of patients do not respond to standard medical and surgical treatment, thus continuously increasing the symptomatologic and socio-economic burden of this disease.

Hypothesis: The investigators believe that the addition of azithromycin (AZI) to the treatment regimen of patients with refractory CRS failing conventional medico-surgical treatment will be beneficial in a symptomatologic and endoscopic level.

Primary objective: 1- To evaluate whether Azithromycine 250 mg PO three times weekly is effective in controlling signs and symptoms of CRS in high-risk patients unresponsive to standard management after endoscopic sinus surgery (ESS) with budesonide irrigations.

Secondary objectives:

i) Validate a simple and concise treatment algorithm for patients refractory to standard CRS treatment of ESS and BUDI, with the addition of low-dose AZI.

ii) Characterise and define the population deemed "high-risk" for standard CRS treatment failure by evaluating: 1) demographics, 2) inflammatory states and 3) the nasal flora microbiome of patients at the different follow-up points of this study.

iii) Explore the mechanisms of AZI by assessing the changes in inflammatory states and the nasal flora microbiome associated with successful AZI therapy.

Methods: Inclusion of all patients admitted for endoscopic sinus surgery (ESS) for CRS operated by the same surgeon (MD). Following their first postoperative visit (2 weeks), all patients will receive nasal irrigations with budesonide (BUDI) twice daily for 4 months and will be re-evaluated. If there is a failure of treatment, patients eligible to receive AZI will be randomized in to two groups, AZI 250mg or a placebo three times a week for 4 months. At every follow-up, complete endoscopic exams will be performed, along with sinus cultures and brush cytology.

Population: All patients deemed "high-risk" with CRS admitted for ESS between October 2014 and October 2015.

ELIGIBILITY:
Inclusion Criteria:

Patients with ≥1 of the following criteria:

* history of sinus surgery,
* first sinus surgery at ≤38 years of age,
* an absolute eosinophilia of ≥500 cells/mm,
* serum IgE levels of >150 kIU/L,
* a Gram negative bacteria in a sinus culture,
* the presence of intra-operative eosinophilic mucin.

Exclusion Criteria:

* Patients with cystic fibrosis, inverted papillomas, osteomata, mucoceles or other lesions of the base of skull will be excluded.
* Patients with an elevated cardiovascular disease risk will be excluded from the randomized clinical trial part of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 129 (Actual)
Dates: Start 2014-11 (Actual); Primary Completion 2017-08-15 (Actual); Study Completion 2017-12-31 (Actual)

PRIMARY OUTCOMES:
Signs and symptoms outcome to Azithromycin | 4 months
  Evaluate if Azithromycin 250mg by mouth, three times a week for four months will be effective in controlling signs and symptoms of chronic rhinosinusitis patients at a high-risk of recurrence following standard medical and surgical treatment. Disease level is evaluated through nasal endoscopy.

SECONDARY OUTCOMES:
Treatment algorithm validation | 8 months
  Validate a simple and concise treatment algorithm for patients refractory to standard CRS treatment of ESS and BUDI, with the addition of low-dose AZI.
High-risk population | 12 months
  Characterise and define the population deemed "high-risk" for standard CRS treatment failure by evaluating:
  1. The demographics of this population
  2. The inflammatory state of patients at the different follow-ups (serum biomarkers)
  3. The microbiome of the nasal flora of patients at the different follow-ups (microbial cultures)
Azithromycin mechanism of action | 12 months
  Explore the mechanisms of action of AZI by assessing the changes in inflammatory states (serum biomarkers and epithelium inflammation) and the nasal flora microbiome (microbial cultures) associated with successful AZI therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Y Desrosiers, MD, FRCSC, Principal Investigator — CHUM
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

REFERENCES:
- [Background] Maniakas A, Desrosiers M. Azithromycin add-on therapy in high-risk postendoscopic sinus surgery patients failing corticosteroid irrigations: A clinical practice audit. Am J Rhinol Allergy. 2014 Mar-Apr;28(2):151-5. doi: 10.2500/ajra.2013.27.4017. Epub 2013 Dec 13. PMID 24598145
- [Background] Desrosiers MY, Kilty SJ. Treatment alternatives for chronic rhinosinusitis persisting after ESS: what to do when antibiotics, steroids and surgery fail. Rhinology. 2008 Mar;46(1):3-14. PMID 18444486
- [Background] Desrosiers M, Evans GA, Keith PK, Wright ED, Kaplan A, Bouchard J, Ciavarella A, Doyle PW, Javer AR, Leith ES, Mukherji A, Robert Schellenberg R, Small P, Witterick IJ. Canadian clinical practice guidelines for acute and chronic rhinosinusitis. J Otolaryngol Head Neck Surg. 2011 May;40 Suppl 2:S99-193. English, French. PMID 21658337
- [Background] Nader ME, Abou-Jaoude P, Cabaluna M, Desrosiers M. Using response to a standardized treatment to identify phenotypes for genetic studies of chronic rhinosinusitis. J Otolaryngol Head Neck Surg. 2010 Feb;39(1):69-75. PMID 20122348
- [Derived] Renteria AE, Maniakas A, Pelletier A, Filali-Mouhim A, Brochiero E, Valera FCP, Adam D, Mfuna LE, Desrosiers M. Utilization of Transcriptomic Profiling to Identify Molecular Markers Predicting Successful Recovery Following Endoscopic Sinus Surgery for Chronic Rhinosinusitis. Otolaryngol Head Neck Surg. 2023 Dec;169(6):1662-1673. doi: 10.1002/ohn.482. Epub 2023 Aug 25. PMID 37622488
- [Derived] Renteria AE, Maniakas A, Mfuna LE, Asmar MH, Gonzalez E, Desrosiers M. Low-dose and long-term azithromycin significantly decreases Staphylococcus aureus in the microbiome of refractory CRS patients. Int Forum Allergy Rhinol. 2021 Feb;11(2):93-105. doi: 10.1002/alr.22653. Epub 2020 Jul 26. PMID 32713109